CLINICAL TRIAL: NCT00093314
Title: An Open-labeled, International, Multicenter, Dose Escalating, Phase I/II Trial of HuMax-CD20, a Fully Human Monoclonal Anti-CD20 Antibody, in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Brief Title: HuMax-CD20 in Chronic Lymphocytic Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Acquired asset
Sponsor: GlaxoSmithKline (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hx-CD20-402
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2007-01

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; B-cell Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell | interventions — ofatumumab

INTERVENTIONS:
Drug: HuMax-CD20

SUMMARY:
The purpose of this trial is to determine the safety and efficacy of HuMax-CD20 as a treatment for Chronic Lymphocytic Leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Lymphocytic Leukemia
* Circulating lymphocytes above a specific level
* Circulating lymphocytes showing certain markers

Exclusion Criteria:

* Previous treatment with rituximab or alemtuzumab within 6 months prior to enrollment in study.
* Previous stem cell transplantation.
* Received any of the following treatments within 4 weeks prior to entering this trial: A) Anti-cancer therapy, B) Glucocorticoids unless less than 10 mg per day, C) Radiotherapy.
* HIV positivity.
* Hepatitis B or hepatitis C.
* Other cancerous diseases, except certain skin cancers and cervix cancer.
* Certain serious medical conditions, including kidney or liver disease, some psychiatric illnesses, and stomach, heart, hormonal, nerve or blood diseases.
* Participation in another trial with a different new drug 4 weeks prior to enrollment in study.
* Current participation in any other clinical study.
* Pregnant or breast-feeding women.
* Women of childbearing age who are unable or unwilling to use adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Hospitals and Clinics, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Struemper H, Sale M, Patel BR, Ostergaard M, Osterborg A, Wierda WG, Hagenbeek A, Coiffier B, Jewell RC. Population pharmacokinetics of ofatumumab in patients with chronic lymphocytic leukemia, follicular lymphoma, and rheumatoid arthritis. J Clin Pharmacol. 2014 Jul;54(7):818-27. doi: 10.1002/jcph.268. Epub 2014 Jan 28. PMID 24443277
- [Derived] Coiffier B, Losic N, Ronn BB, Lepretre S, Pedersen LM, Gadeberg O, Frederiksen H, van Oers MH, Wooldridge J, Kloczko J, Holowiecki J, Hellmann A, Walewski J, Robak T, Petersen J. Pharmacokinetics and pharmacokinetic/pharmacodynamic associations of ofatumumab, a human monoclonal CD20 antibody, in patients with relapsed or refractory chronic lymphocytic leukaemia: a phase 1-2 study. Br J Haematol. 2010 Jul;150(1):58-71. doi: 10.1111/j.1365-2141.2010.08193.x. Epub 2010 Apr 16. PMID 20408846
- [Derived] Coiffier B, Lepretre S, Pedersen LM, Gadeberg O, Fredriksen H, van Oers MH, Wooldridge J, Kloczko J, Holowiecki J, Hellmann A, Walewski J, Flensburg M, Petersen J, Robak T. Safety and efficacy of ofatumumab, a fully human monoclonal anti-CD20 antibody, in patients with relapsed or refractory B-cell chronic lymphocytic leukemia: a phase 1-2 study. Blood. 2008 Feb 1;111(3):1094-100. doi: 10.1182/blood-2007-09-111781. Epub 2007 Nov 14. PMID 18003886